CLINICAL TRIAL: NCT00077987
Title: A Phase II Study Of SU011248 In Patients With Metastatic Colorectal Cancer Who Have Previously Failed Treatment With Irinotecan, Oxaliplatin, And A Fluoropyrimidine, With And Without Bevacizumab
Brief Title: Assessment Of Safety And Efficacy Of SU11248 In Patients With Metastatic Colorectal Cancer Who Have Failed Selected Previous Treatments.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181003; NCT00082771 (obsolete NCT alias)
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2005-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sunitinib

INTERVENTIONS:
Drug: SU011248

SUMMARY:
Assessment of safety and efficacy of SU11248 in patients with metastatic colorectal cancer who have failed selected previous treatments.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* Failed selected cancer therapies in the past.

Exclusion Criteria:

* Prior treatment with tyrosine kinase inhibitors or VEGF inhibitors other than bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2003-12; Study Completion 2005-04

PRIMARY OUTCOMES:
Anti-tumor efficacy

SECONDARY OUTCOMES:
Tumor control survival safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer